CLINICAL TRIAL: NCT02944032
Title: Multimodal Intervention Trial for Cognitive Deficits in Neurofibromatosis Type 1: Efficacy of Computerized Cognitive Training and Stimulant Medication
Brief Title: Efficacy of Computerized Cognitive Training and Stimulant Medication in Neurofibromatosis Type 1
Acronym: COGTRAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kristina Hardy (Other)
Collaborators: Children's National Research Institute (Other); Royal Children's Hospital (Other); Children's Hospital Los Angeles (Other); Sydney Children's Hospitals Network (Other)
Responsible Party: Sponsor-Investigator, Kristina Hardy, PhD, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00007343
Record Dates: First submitted 2016-05-25; First posted 2016-10-25 (Estimated); Last update posted 2022-03-03 (Actual); Status verified 2022-03

CONDITIONS: Neurofibromatosis Type 1
MeSH Terms: conditions — Neurofibromatosis 1

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cogmed (Experimental): Cogmed RM is a computer program that consists of twelve visually-engaging and interesting exercises that target skills involving visuo-spatial and verbal Working Memory. During the intervention, children complete 25 training sessions. Children are asked to complete between 3 and 5 sessions per week, so the total treatment time to complete 25 sessions may range from 5 to 9 weeks. For children completing CogmedRM, sessions typically last between 25 and 45 minutes, depending on the child's working memory span.
  Interventions: Other: CogmedRM
- MobyMax (Active Comparator): MobyMax's "Reading Stories" program is a program that focuses on reading comprehension skills. Participants will start their training with stories that are matched to their reading "grade" level. Each grade contains 30 lessons, with 3 stories in each lesson. Participants are given questions to answer at the conclusion of each story, and children advance or remain at that level depending on the progression of their reading skill. Participants randomized to this program will be asked to train 30-45 minutes per session for 25 training sessions over a 5 to 9 week period.
  Interventions: Other: Mobymax

INTERVENTIONS:
Other: CogmedRM — Cogmed RM is a computer program that consists of twelve visually-engaging and interesting exercises that target skills involving visuo-spatial and verbal Working Memory. Difficulty of the tasks is automatically adjusted on a trial-by-trial basis throughout each training session to match a child's current working memory span, such that as the child becomes more proficient, the exercises become more difficult. During the intervention, children complete 25 training sessions. Children are asked to complete between 3 and 5 sessions per week, so the total treatment time to complete 25 sessions may range from 5 to 9 weeks. For children completing CogmedRM, sessions typically last between 25 and 45 minutes, depending on the child's working memory span.
  Arms: Cogmed
Other: Mobymax — MobyMax's "Reading Stories" program is a program that focuses on reading comprehension skills. Participants will start their training with stories that are matched to their reading "grade" level. Each grade contains 30 lessons, with 3 stories in each lesson. Participants are given questions to answer at the conclusion of each story, and children advance or remain at that level depending on the progression of their reading skill. Participants randomized to this program will be asked to train 30-45 minutes per session for 25 training sessions over a 5 to 9 week period.
  Arms: MobyMax

SUMMARY:
The main objective of the study is to assess the efficacy of a home-based, computerized cognitive training (CT) program, called CogmedRM, targeted to improve working memory in children with NF1 and working memory difficulties. This is a Phase II randomized parallel group controlled clinical trial comparing two interventions on cognitive outcomes. Participants will be stratified by stimulant medication use and randomized equally between the two interventions within stratum. Participants will be in the study for to 11 weeks.

DETAILED DESCRIPTION:
Cognitive deficits are the most important cause of long-term dysfunction in patients with Neurofibromatosis type 1 (NF1). Among the most frequently-occurring difficulties are problems with attention, working memory (WM), and executive functioning (EF). Remediation and interventions to improve those deficits have the potential to impact the quality of life and long-term prognosis in this population. Cognitive training (CT) programs have increasingly been used independently or in conjunction with pharmacotherapies in children with accidental or disease-related brain injury. CogmedRM is both the most well-researched and widely-used CT program for remediation of WM deficits. Results from numerous randomized, controlled trials conducted with a variety of pediatric and adult patient populations generally show that CogmedRM training is associated with robust gains in performance-based WM scores over the short term, with some variability in improvement across disease groups. A single arm pilot study of CogmedRM in a sample of children with NF1 conducted at Children's National Medical Center has shown that the approach is likely feasible and acceptable to families.

Because many children with NF1 are treated with stimulant medications, and there is biological evidence that both CT and Methylphenidate act on dopaminergic systems, the investigators are also interested in examining whether or not there is a synergistic effect between these widely available and safe interventions. Thus, the aim is to assess the efficacy of a home-based, computerized cognitive training (CT) program in a sample of 90 children aged 8-16 with NF1 and working memory difficulties. This study will be conducted over the span of four years. If the participant qualifies following baseline testing, he/she will be randomized to the intervention, CogmedRM, or the active control condition, MobyMax (an online reading program). The participant will have 5-9 weeks to complete the program and will have follow-up testing 2 weeks after finishing the program. If CT, either singly or in combination with stimulant medication, can be shown to be efficacious in a sample of NF1 pediatric patients at high risk for neurocognitive deficits, this intervention plan could be rapidly translated to clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. 8-16 years old at time of screening
2. NF1 Diagnosis based on National Institute of Health (NIH) criteria
3. Has an identified caregiver who is willing and able to oversee the training practice during the intervention period
4. Has access to a telephone and phone number where they can be reached
5. Both patient and caregiver have reading, speaking, and listening comprehension of English
6. Treated with a stable dose of stimulant medication for at least the last 30 days and not planning to change the dose during study participation or receiving no stimulant medications for at least the last 30 days and not planning to initiate a trial of stimulant medications for the duration of the study.
7. >1 Standard Deviation (SD) below the mean on the WISC-V-Integrated Spatial Span Backwards task or a Spatial Span Backwards score >1 SD below the participant's estimated IQ.

Exclusion Criteria:

1. Full scale IQ<70, as estimated by WASI-II (Block Design, Vocabulary, Matrix Reasoning, Similarities).

   Note: In cases where there is a statistically significant difference between verbal IQ and performance IQ (.05 level as determined by the WASI-II manual), participants will be eligible if at least one of these quotients is 70 or above
2. Current treatment for intracranial lesions, progressive tumors as per MRI evaluation or treatment with chemotherapy within the past 6 months
3. A motor, visual, or auditory handicap that prevents computer use

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 103 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
Change in CogState One-back subtest | From baseline to end of training, up to 11 weeks
  Computerized task of working memory

SECONDARY OUTCOMES:
Change in Attention Deficit Hyperactive Disorder- Rating Scale | From baseline to end of training, up to 11 weeks
  Parent-completed rating scale
Change in Wechsler Intelligence Scale for Children-Fifth Edition-Integrated Spatial Span Backward | From baseline to end of training, up to 11 weeks
  Visual-spatial working memory task
Change in Wechsler Intelligence Scale for Children-Fifth Edition-Integrated Digit Span Backward | From baseline to end of training, up to 11 weeks
  Auditory working memory task
CogState One-card Learning | From baseline to end of training, up to 11 weeks
  Computerized attention and executive functioning tasks
Change in Behavior Rating Inventory of Executive Functioning (BRIEF) Working Memory Index | From baseline to end of training, up to 11 weeks
  Parent-completed questionnaire
Change in Test of Word Reading Efficiency-Second Edition (TOWRE-2) Scores | From baseline to end of training, up to 11 weeks
  Child-completed reading task
Change in Test of Everyday Reading Comprehension (TERC) Scores | From baseline to end of training, up to 11 weeks
  Child-completed reading task
Change in Behavior Rating Inventory of Executive Functioning (BRIEF) Metacognition Index | From baseline to end of training, up to 11 weeks
  Parent-completed questionnaire
CogState Groton Maze Learning Task | From baseline to end of training, up to 11 weeks
  Computerized task of executive functioning
Change in Wechsler Intelligence Scale for Children-Fifth Edition-Integrated Letter-Number Sequencing | From baseline to end of training, up to 11 weeks
  Auditory working memory task

CONTACTS AND LOCATIONS:
Overall Officials: Kristina Hardy, PhD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Health System, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-10): https://cdn.clinicaltrials.gov/large-docs/32/NCT02944032/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-21): https://cdn.clinicaltrials.gov/large-docs/32/NCT02944032/ICF_001.pdf